CLINICAL TRIAL: NCT05255029
Title: Clinical Investigation of the Monofocal Toric IOL POD T 49P in Cataractous Eyes
Brief Title: Clinical Investigation of a Monofocal Toric Intra Ocular Lens (IOL) in Cataractous Eyes
Acronym: PHY2107
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beaver-Visitec International, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHY2107
Record Dates: First submitted 2021-11-26; First posted 2022-02-24 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Cataract; Lens Opacities; Astigmatism
Keywords: Intraocular Lens; Monofocal; Toric Lens
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Intervention Model Description: 1) Summary of investigational lens Model: POD T 49P General name: PODEYE Toric Construction Single-piece construction lens consisting of the optic and the haptic made of the same material, optic diameter: 6.0 mm, overall length: 11.4 mm (Fig.1). Cylinder power is added on the posterior optics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PODEYE Toric Intra Ocular Lens Implantation experimental (Experimental): Implantation of PODEYE toric intraocular lenses.
  Interventions: Device: POD T 49P implantation experimental

INTERVENTIONS:
Device: POD T 49P implantation experimental — The investigational lens will be implanted within the capsular bag after removal of the natural crystalline lens following phacoemulsification and alignment the toric axis of investigational lens to the intend axis which was calculated by the Toric calculator software. When enroll the test lenses into both eyes, the lens is implanted first to the eye with more advanced cataract. If both eyes have a similar degree of cataract, perform the surgery first for the right eye. The timing of surgery the investigational lens into the fellow eye will be determined after the investigator and the investigator (hereinafter referred to as the investigator) have confirmed the safety of the previously operated eye.

SUMMARY:
This is a Multi-center, single-arm and non-masked study whereby patients undergoing routine cataract surgery be implanted with a hydrophobic acrylic monofocal toric intraocular lens PODEYE TORIC (model POD T 49P).

DETAILED DESCRIPTION:
This is a Multi-center, single-arm and non-masked study whereby patients undergoing routine cataract surgery will be implanted with a hydrophobic acrylic monofocal toric intraocular lens PODEYE TORIC. The device under investigation is a hydrophobic acrylic monofocal toric intraocular lens (IOL) manufactured by the sponsor of this study (BVI Medical). The refractive power of the lens has a spherical and a cylindrical component. The IOLs will be implanted in the course of routine cataract surgery and will benefit to patients suffering from cataract development and showing pre-existing corneal astigmatism.

In total approx. 28 patients, 56 eyes will be recruited for this clinical study and undergo implantation of PODEYE TORIC intraocular lens.

Subjects participating in the trial will attend a total of maximum 6 study visits over a period of 120-180 days (preoperative, operative, 1-2 days, 7-14 days, 30-60 days, 120-180 days, postoperative visits). Subjects would have the option for unscheduled visits if required medically.

ELIGIBILITY:
The patient who meets all criteria specified in the following 1) through 8)

1. Adults, 20 years of age or older at the time of informed consent, of either gender, diagnosed with cataract;
2. Able to comprehend and sign a statement of informed consent;
3. Willing and able to complete all required postoperative visits;
4. Calculated lens power within the available range;
5. Subject with corneal astigmatism or subjects who is judged by the investigator or investigator to correct of astigmatism as a result of considering the predicted surgical induced astigmatism.
6. Planned cataract removal by phacoemulsification;
7. Target postoperative refraction is emmetropia and potential postoperative Collected Distance Visual Acuity (CDVA) of 0.5 decimal or better in both eyes;
8. Clear intraocular media other than cataract in both eyes;

[Justification for the inclusion criteria]

1 and 6: Cataract extraction is the indication of the clinical study. 2 and 3: One of GCP requirements 4 and 5: Essential condition for implant of the investigational lens. 7 and 8: Conditions to minimize the potential non-IOL factors which may affect the visual acuity data

(3) Exclusion Criteria [Exclusion Criteria Prior to Surgery] The patient who meets any criteria specified in the following 1) through 20).

1. Subjects with diseases that affect postoperative visual acuity in the cornea (keratitis, corneal degeneration, corneal dilatation, corneal edema);
2. Previous corneal transplant;
3. Previous refractive surgery;
4. Irregular corneal aberration
5. Subjects with diseases that affect postoperative visual acuity in the retina (retinal degeneration, diabetic retinopathy, retinal detachment);
6. Poor mydriasis;
7. Glaucoma or ocular hypertension;
8. Optic nerve atrophy;
9. Extremely shallow anterior chamber;
10. Aniridia;
11. Iris neovascularization;
12. Microphthalmos;
13. Amblyopia;
14. Rubella, atopic or traumatic cataract;
15. Recurrent severe anterior or posterior segment inflammation of unknown etiology;
16. Subjects who may be expected to require ocular surgery during this study;
17. The axial length cannot be measured with an optical biometry;
18. Pregnancy, lactating or possible pregnant;
19. Participation in any clinical study (drug or device) within 3 months prior to participating this study, planned participation another clinical study during this study, or currently participating in another study.
20. Disqualified by the investigator or the sub-investigator because of physical or ophthalmic diseases

[Exclusion Criteria During Surgery] The patient who meets any criteria specified in the following 1) through 8).

1. Mechanical or surgical manipulation required to enlarge the pupil;
2. Excessive iris mobility;
3. Uncontrollable intraocular pressure;
4. Continuous Curvilinear Capsulorrhexis (CCC) with incomplete circle or tear;
5. Zonular or capsular rupture or tear;
6. Significant anterior chamber hyphema;
7. Significant vitreous loss;
8. IOL could not be fixed in the lens capsule;

In the event of zonular damage, capsulorhexis tear, or decentered capsulorhexis during surgery, the surgeon should decide whether the stability of the Intra Ocular Lens (IOL) would be compromised by the complication. If the IOL stability would be compromised, the investigational IOL should not be implanted, the subject should be discontinued from the study, and the surgeon should make arrangements to implant an alternative non-investigational IOL.

[Justifications for the exclusion criteria] {Exclusion Criteria Prior to Surgery} 1, 2, 3, 4, 5, 7, 8, 14, 15, 16 and 20: Factors potentially affecting effectiveness evaluability and criteria to secure safety of study subjects 6, 13 and17: Factors potentially affecting effectiveness evaluability 9, 10, 11, 12, 18 and 19: Criteria to secure safety of study subjects

{Exclusion Criteria During Surgery}

1, 2, 4, 5 and 8: Factors potentially affecting effectiveness evaluability 3, 6 and 7: Criteria to secure safety of study subjects

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-12-24 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Uncorrected visual acuity at Visit 4 | Postoperative Day 120-180
  Uncorrected visual acuity at 5 m will be measured. Convert decimal visual acuity to logMAR value using the following formula.
  logMAR value = log10 (1/decimal visual acuity)
Amount of astigmatism at Visit 4 | Postoperative Day 120-180
  Manifest cylindrical refraction for Best Collected Distance Visual Acuity will be measured at Visit 4.

SECONDARY OUTCOMES:
Best Corrected Distance Visual Acuity | Pre-Op, 1 week postoperative, 1 month postoperative, 6 months postoperative.
  Best Corrected Distance Visual Acuity at 5 m will be measured. The objective is to compare CDVA above defined thresholds of the investigational product.
Manifest cylindrical refraction | Pre-Op, 1 month postoperative, 6 months postoperative
  Manifest cylindrical refraction for Best Collected Distance Visual Acuity will be measured.
IOL rotation | Pre-Op, 1 month postoperative, 6 months postoperative
  After mydriasis, a photograph of the anterior segment of the test lens is taken using an anterior segment analyzer, and the angle of the toric mark with respect to the horizon is measured as the axial angle. Calculate the number of the eye and the percentage of less than 5 degrees, more than 5 degrees to less than 10 degrees, more than 10 degrees to less than 20 degrees.

OTHER OUTCOMES:
Intraocular pressure (IOP) measurement | Pre-Op, 1 day postoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative
  The IOP will be measured with non-contact tonometer as part of the routine follow up examinations. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
Slitlamp examination - Corneal Status | Pre-Op, 1 day postoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Corneal Status
Fundus examination with dilated pupil | Pre-Op, 1 day postoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Fundus
Slitlamp examination | Pre-Op, 1 day postoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  * Signs of inflammation
  * Anterior chamber cells,
  * Anterior chamber flare,
  * Cystoid macular oedema,
  * Hypopyon, and
  * Endophthalmitis
Slitlamp examination - Retinal detachment | Pre-Op, 1 day postoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative, 24 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Retinal detachment
Slitlamp examination - IOL decentration | 1 day postoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative, 24 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • IOL decentration
Slitlamp examination - IOL tilt | 1 day postoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • IOL tilt
Adverse events | Pre-Op, during surgery, 1 day postoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative
  Record the presence or absence of AE after Informed Consent.
Device deficiencies | Pre-Op, during surgery, 1 day postoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative
  Record the presence or absence of device deficiencies after Informed Consent.

CONTACTS AND LOCATIONS:
Overall Officials: MIYATA Kazunori, MD, Principal Investigator — Miyata Eye Hospital
Locations (4):
- Japan (4):
  - Chukyo Eye Clinic, Nagoya, Aichi-ken
  - Roppongi Shiba Eye Clinic, Minato-Ku, Tokyo
  - Miyata Eye Hospital, Miyazaki
  - Fujita Eye Clinic, Tokushima

IPD SHARING:
Plan to Share IPD: No